CLINICAL TRIAL: NCT05965284
Title: A Prospective, Open-label, Controlled, Single Center Clinical Study of the Efficacy and Safety for Telitacicept in the Remission Maintenance Treatment of ANCA-associated Vasculitis
Brief Title: Efficacy and Safety for Telitacicept in the Remission Maintenance Treatment of ANCA-associated Vasculitis (TTCAZAREM)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR-K2374
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: ANCA-associated Vasculitis; Maintenance Therapy
Keywords: ANCA-associated Vasculitis; Telitacicept; Azathioprine; Relapse rate
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Azathioprine; telitacicept

STUDY DESIGN:
Intervention Model Description: prospective, randomized, open-label, control, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azathioprine treatment arm (Other): Patients will be treated with Azathioprine 100mg per day for 12 months combined with prednisone no more than 10mg daily. The dosage of prednisone is tapered in the study period while sustained remission achieved. All included patients will be treated with TMPco 2 tablets per day during the study period if not contraindicated or intolerant.
  Interventions: Drug: Azathioprine
- Telitacicept treatment arm (Experimental): Patients will be treated with Telitacicept 160mg per week combined with Azathioprine 100mg per day for 12 months combined with prednisone no more than 10mg daily. The dosage of prednisone is tapered in the study period while sustained remission achieved. All included patients will be treated with TMPco 2 tablets per day during the study period if not contraindicated or intolerant.
  Interventions: Drug: Azathioprine; Drug: Telitacicept

INTERVENTIONS:
Drug: Azathioprine — All patients included into this study will be treated with Azathioprine tablets 100mg QD for 12 months.
Drug: Telitacicept — Patient will be treated with Telitacicept (Taiai the commercial name) 160 mg every week subcutaneously for 12 months
  Other Names: Taiai for commercial name
  Arms: Telitacicept treatment arm

SUMMARY:
This study is a prospective, open-labelled, randomized, controlled, single-center clinical trial. The aim of this study is to compare the remission rate of patients treated with Telitacicept combined with azathioprine and azathioprine alone in remission-maintenance treatment of AAV.

DETAILED DESCRIPTION:
Background: The basic theme of AAV is relapse and remission. The maintenance therapy of AAV aimed to reduce or prevent relapse is very challenge. Although many medications have been used for the maintenance of AAV, Telitacicept (a BAFF/APRIL dual-target-inhibitor, which has been proved to be effect in treatment of SLE) has not been studied yet. One study tested the efficacy of Belimumab in the maintenance therapy for AAV. When taken Rituximab as remission-induction treatment, no relapse was observed. However, the sample size of this study is small, and the Belimumab, as a BAFF inhibitor, was not been proved to have effect on APRIL.

Many experiences have been accumulated about the efficacy and safety of Telitacicept in Chinese patients with rheumatic diseases. But there is no study to show its effectiveness in the reduction of the relapse of AAV in China. In this study, we add Telitacicept to azathioprine in maintain treatment in AAV patients who receive Rituximab as remission-induction treatment, to compare the relapse rates of Telitacicept combining azathioprine and azathioprine alone in maintenance therapy of AAV.

Objectives: To compare the relapse rates of Telitacicept combining azathioprine and azathioprine alone in maintenance treatment of AAV.

Study Design: This is a prospective, randomized, open-label, control, pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 65 years, both genders can be included.
2. Patients who are newly diagnosed or relapsing granulomatosis with polyangiitis or microscopic polyangiitis must fulfill the 2022 ACR/EULAR classification criteria of GPA or MPA.
3. Patients who are in complete remission after combined treatment with glucocorticoids and Rituximab. Remission is defined as a Birmingham Vasculitis Activity Score (BVAS version 3) of 0. And the daily dosage of prednisone are no more than 10mg (or equivalent).
4. Patients have to be ANCA-positive at diagnosis or during the course of their disease.

Exclusion Criteria:

1. Patients with TPMT gene mutation.
2. Patients who had been treated with either AZA but relapsed in the past.
3. Patients who had been treated with either AZA but had to stop due to adverse events or intolerance.
4. Patients who have planned for pregnancy in next 1.5 years.
5. Patients with severe liver dysfunction(defined as the 2-folds elevation of normal upper limit or Child grade III), heart failure or ESRD(eGFR<30ml/min).
6. Patients with uncontrolled sever hypertension, diabetes, active bacteria or fungal infection;
7. Patients with active hepatitis virus infection as well as patients who have active mycobacteria infection;
8. Patients who had other autoimmune diseases.
9. Patients with malignancy.
10. Patients who are not eligible according to the judge of the principal investigators or site investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The time of first relapse during 12 months follow-up of two groups | from inclusion to the end of the study, 12 months in total
  The time from baseline to first relapse(re-appearance of disease with a BVAS >0) of patients during 12 months follow-up of two groups

SECONDARY OUTCOMES:
The percentage of patients with severe relapse at months 12 | from inclusion to the end of the study, 12 months in total
  The percentage of patients with severe relapse (re-appearance or worsening of disease with a BVAS ≥6 and involvement of at least one major organ, a life-threatening manifestation, or both) at months 12
The percentage of patients with moderate relapse at months 12 | from inclusion to the end of the study, 12 months in total
  The percentage of patients with moderate relapse (re-appearance or worsening of disease with a BVAS ≥3 without involvement of major organ or life-threatening manifestation) at months 12
The percentage of patients with mild relapse at months 12 | from inclusion to the end of the study, 12 months in total
  The percentage of patients with mild relapse (re-appearance or worsening of disease with a 0 < BVAS < 3 without involvement of major organ or life-threatening manifestation) at months 12
The percentage of patients with sustained remission at months 12 | from inclusion to the end of the study, 12 months in total
  The percentage of patients with sustained remission (BVAS =0 without dosage increase of glucocorticoid) at months 12
The rate of adverse events | from inclusion to the end of the study, 12 months in total
  The rate of adverse events and their severity (Severe events were defined as the adverse events of grade 3 or 4, deaths caused by any cause, cancers, side effects that necessitate hospitalization) in both two groups during the study period.
The percentage of patients who progress to ESRD | from inclusion to the end of the study, 12 months in total
  The percentage of patients who progress to ESRD at the end of the study
The rate of complication of AAV | from inclusion to the end of the study, 12 months in total
  The rate of complication of AAV in both treatment groups during 12 months of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: JIng Li, M.D., Principal Investigator — Peking Unione Mdecial College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China